CLINICAL TRIAL: NCT05333666
Title: The Association Between Non-vitamin K Antagonist Oral Anticoagulant Concentration and Clinical Outcomes (The Direct Oral AntiCoagulant Registry in Taiwan, DOACT)
Brief Title: The Association Between Non-vitamin K Antagonist Oral Anticoagulant Concentration and Clinical Outcomes.
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202201014RINB
Record Dates: First submitted 2022-03-15; First posted 2022-04-19 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Age over 20 years and under non-vitamin K antagonist oral anticoagulant therapy
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — This investigation aims to collect and analyze the data from a cohort. During the cohort development, all participants received venous puncturing for NOAC concentration measurement. However, the standard treatment protocol was not changed after study enrollment. In this retrospective cohort study, we only collect data from the cohort without further intervention to the participants.

SUMMARY:
Introduction: Non-vitamin K antagonist oral anticoagulants (NOAC) is the first line therapy to prevent ischemic stroke or systemic thromboembolism among atrial fibrillation (AF) patients. Since 2016, our study team enrolled patients under NOAC therapy in National Taiwan University Hospital, and measured their NOAC concentration to develop a cohort of NOAC treatment and NOAC concentration.

Study purpose: Based on the cohort of NOAC therapy, we aim to investigate factors driving high or low NOAC concentration, and link NOAC concentration to clinical outcomes.

Methods: For all the participants in the cohort, we will retrieve their basic characteristic, concurrent medications, laboratory tests and clinical outcomes such as ischemic stroke, systemic thromboembolism, intracranial hemorrhage, major bleeding and death from the electronic medical records. The NOAC concentration will be compared to the expected range reported in clinical trials to define higher, within or lower than expected range. Univariate logistic regression will be used first, followed by multivariate logistic regression to investigate factors associated with high or low NOAC concentration. The relationship between NOAC concentration and clinical outcomes will be investigated by using the Cox proportional hazard model.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 20 years.
* Under NOAC therapy.

Exclusion Criteria:

* Failed to provide at least one blood sample for NOAC concentration measurement.
* Declined to provide informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under NOAC therapy.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with ischemic stroke, transient ischemic attack or systemic thromboembolism. | From the date of study enrollment to end of NOAC exposure, death, occurrence of aforementioned outcome (ischemic stroke, transient ischemic attack or systemic thromboembolism) or end of the study, whichever comes first, assessed up to 100 months.
  ischemic stroke, defined as an episode of neurological dysfunction caused by focal cerebral infarction. Transient ischemic attack is defined as a transient episode of neurological dysfunction caused by focal brain ischemia without acute infarction. The diagnose tool included clinical and radiological diagnosis included CT and MRI. Systemic thromboembolism includes myocardial infarction, venous thromboembolism, coronary artery disease or peripheral arterial occlusive disease.

SECONDARY OUTCOMES:
Major or life-threatening bleeding | From the date of study enrollment to end of NOAC exposure, death, occurrence of major bleeding or life-threatening bleeding classified by using the PLATO criteria or end of the study, whichever comes first, assessed up to 100 months
  The severity of bleeding is classified by using the PLATO criteria

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei, Please Select
  - National Taiwan University Hospital, Taipei